CLINICAL TRIAL: NCT01690039
Title: Comparison of Furosemide/Fludrocortisone With Ammonium Chloride Loading Test in the Diagnosis of Incomplete dRTA in Kidney Stone Formers
Brief Title: Influence of Polymorphisms in the ATP6V1 Gene of the V-ATPase on the Development of Incomplete Distal Renal Tubular Acidosis
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 090/12
Record Dates: First submitted 2012-09-10; First posted 2012-09-21 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Acidosis, Renal Tubular; Nephrolithiasis; Vacuolar Proton-Translocating ATPases
Keywords: renal tubular acidosis; V-ATPase; kidney stones
MeSH Terms: conditions — Acidosis, Renal Tubular; Nephrolithiasis; Kidney Calculi | interventions — Furosemide; Fludrocortisone; fludrocortisone acetate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All study participants: Furosemide-Fludrocortisone-Test and Ammonium chloride-Loading Test will be performed in renal stone patients.
  Interventions: Drug: Furosemide-Fludrocortisone-Test (test for urinary acidification)

INTERVENTIONS:
Drug: Furosemide-Fludrocortisone-Test (test for urinary acidification) — The presence of a lack of urinary acidification will be assessed by an appropriate test in all patients.
  Other Names: Application of Furosemide (Lasix® ) and Fludrocortisone (Florinef®)

SUMMARY:
Purpose

1. To compare the performance of the two currently employed urinary acidifications tests in stone formers, the furosemide/fludrocortisone and ammonium chloride loading test.
2. To study the impact of polymorphisms in the genes ATP6V1B1, ATP6V0A4 and SLC4A1 on urinary acidification in stone formers.

ELIGIBILITY:
Inclusion Criteria:

* One or more episodes of nephrolithiasis

Exclusion Criteria:

* Absence of informed consent
* All conditions affecting renal acidification
* Pregnancy
* Nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffered from at least one kidney stone episode.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12-31 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Capability of urinary acidification | Five to six hours

SECONDARY OUTCOMES:
Polymorphisms in the ATP6V1 gene | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Fuster, Attending physician Nephrology, Principal Investigator — Department of Nephrology and Hypertension, Bern University Hospital
Locations (1):
- Department of Nephrology and Hypertension, Bern University Hospital, Bern, Switzerland

REFERENCES:
- See also: Institution homepage — http://www.nephrologie.insel.ch/